CLINICAL TRIAL: NCT06037460
Title: TocilizuMab discontinuAtion in GIant Cell Arteritis
Acronym: MAGICA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAMSON PHRCN 2021
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gradual discontinuation of TCZ (Experimental)
  Interventions: Drug: Tocilizumab treatment; Other: questionnaires; Biological: Blood samples; Procedure: 18FDG PET scan
- Immediate discontinuation of TCZ (Active Comparator)
  Interventions: Other: questionnaires; Biological: Blood samples; Procedure: 18FDG PET scan

INTERVENTIONS:
Drug: Tocilizumab treatment — * 1 injection/2 weeks from W0 to W12: W0, W2, W4, W6, W8, W10, W12
  * Then 1 injection/4 weeks until W24: W16, W20, W24
  Arms: Gradual discontinuation of TCZ
Other: questionnaires — HAQ, SF-36, FACIT-Fatigue score
Biological: Blood samples — Additionnal blood samples for immunomonitoring
Procedure: 18FDG PET scan — PETVAS calculation (to be performed between W0 and W8) (optional).

SUMMARY:
Giant cell arteritis (GCA) is a large-vessel vasculitis that typically occurs in people over the age of 50.

Corticosteroids (GC) are the cornerstone of treatment for GCA. French guidelines recommend starting at 0.7 or 1 mg/kg/day at diagnosis, depending on the occurence of ischemic complication(s). Then, it is recommended to gradually decrease their dose to achieve withdrawal in 12 to 24 months.

Despite this treatment, 47% of patients relapse. Relapses are favored by rapid reduction of corticosteroid doses and large vessel involvement at diagnosis. Fortunately, relapses are severe in only 3.3% of cases and ischemic complications are very rare. However, this contributes to prolonging the duration of corticosteroid treatment and thus the risk of cortico-induced adverse events, which have not been significantly reduced in the last 20 years. The main risk factors for the development of steroid-related complications are advanced age and cumulative steroid dose.

For this reason, the development of cortisone-sparing strategies is necessary to improve the management of patients with GCA. Thanks to major advances in the understanding of the pathophysiological mechanisms of GCA, new therapeutic targets have been discovered. For example, the efficacy of tocilizumab (TCZ), an anti-IL-6 receptor monoclonal antibody, has been demonstrated in two phase 2 trials and one phase 3 trial, leading to its approval for the management of patients requiring rapid reduction in corticosteroid doses and/or those relapsing repeatedly on prednisone >7.5 mg/day. In recently published US guidelines, TCZ can even be used at diagnosis to reduce the need for corticosteroid therapy.5 Indeed, TCZ appears to be remarkably effective in controlling GCA activity and saves approximately 2000 mg of prednisone in cumulative dose.

At present, the place of TCZ compared to methotrexate in the therapeutic strategy is still being evaluated, notably through the METOGiA study (PHRC-N 2017), which is being conducted by our team. Inclusions for METOGiA ended in March 2023 with results expected in 2025. Outside of this study, approximately 1500 patients are currently receiving TCZ treatment for GCA (data from ROCHE-CHUGAI).

There is no doubt that TCZ treatment is effective and rather well tolerated in the elderly population, but it generates problems that are not solved to date:

* the cost (~900€/month)
* the difficulty monitoring these patients because the biological markers usually used to monitor GCA (CRP, ESR, fibrinogen) can no longer be measured since TCZ blocks their production by the hepatocytes. Monitoring of disease activity therefore requires very careful clinical examination and the use of expensive imaging tests such as PET scans because GCA can be active despite normal ESR, CRP and fibrinogen levels. Some studies suggest that monitoring serum IL-6 may help identify patients with active disease, but this test is not readily available and the threshold above which relapse should be suspected is unclear because TCZ induces an increase in serum IL-6 levels by blocking IL-6 receptors, even in patients in remission.
* For the same reasons, infections are difficult to detect in patients treated with TCZ.

This raises the question of how to discontinue this treatment, especially since other treatments that do not interfere with CRP, ESR, or fibrinogen measurements are being evaluated.

This shows that this treatment tends to be prolonged well beyond one year when the disease is often in remission without corticosteroids. This is probably related to two factors: 1/ the fear of relapse after treatment withdrawal; 2/ the absence of a scheme for withdrawing TCZ.

The risk of relapse after stopping TCZ has been reported in several studies, in particular the long-term follow-up of phase 2 and 3 trials that demonstrated the efficacy of TCZ for the treatment of GCA. Overall, regardless of the duration of TCZ treatment, the risk of relapse is approximately 40% 6 months after the last injection of TCZ, and the risk of relapse is higher if the large arteries (aorta and its branches) are involved.

Thus, although the available data are limited, it appears that tapering rather than immediately stopping TCZ limits the risk of relapse after full withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* Diagnosis of GCA, defined by the following criteria:

  * Age ≥50 years at diagnosis
  * AND History of ESR ≥50 mm/h OR CRP ≥20 mg/L (optional criterion if temporal artery biopsy (TAB) is positive).
  * AND at least one of the following clinical criteria:

    * At least one unequivocal sign of GCA (recent headache, scalp hyperesthesia, jaw claudication, temporal artery abnormality, visual disturbances of ischemic origin)
    * Clinical sign(s) of polymyalgia rheumatica (PR)
  * AND at least one of the following criteria during GCA follow-up:

    * TAB consistent with the diagnosis of GCA (non-necrotizing vasculitis with a mononuclear cell-rich inflammatory infiltrate or presence of granulomas, with or without multinuclear giant cells)
    * Evidence of temporal artery vasculitis by echo-Doppler of the temporal arteries (unilateral or bilateral halo sign)
    * Evidence of vasculitis of at least one large vessel by imaging:
  * angio-CT or angio-MRI: arterial wall thickening (≥2mm for aorta; ≥1mm for supra-aortic trunks and upper extremity arteries, ≥0.6mm for the cephalic artery, …) and/or T1-weighted contrast.
  * PET: grade 2 or 3* hypermetabolism of the wall of at least one large vessel (aorta, supra-aortic trunks, cephalic vessels, upper extremity arteries) (*i.e., arterial SUVmax ≥ liver SUVmax)
* GCA in remission for at least 12 weeks before randomisation (remission = absence of symptoms due to GCA AND CRP ≤10 mg/L)
* TCZ treatment (IV or SC) or biosimilar initiated 12 to 36 months prior to randomization
* TCZ treatment (IV or SC) or biosimilar not interrupted more than 12 weeks in the 12 months prior to randomization
* Treatment with subcutaneous TCZ (162 mg/week) or biosimilar for at least 12 consecutive weeks prior to randomization
* Treatment with corticoids stopped at least 12 weeks before randomization (hydrocortisone treatment ≤20 mg/day is possible if given at a stable dose for the duration of the study)
* Biological workup dating from less than 6 weeks on the day of randomization, showing good tolerance of tocilizumab:

  * AST and ALT < 1.5 x upper limit of normal (ULN)
  * Hemoglobin >8 g/dL
  * Platelets >100 G/L
  * Neutrophils >1 G/L
  * Lymphocytes >0.5 G/L

Exclusion Criteria:

* Person who is not affiliated with the national health insurance system
* Person subject to a measure of legal protection (guardianship, tutorship)
* Person subject to a court order
* Patient unable to give consent
* Person who does not speak French
* Pre-menopausal women (menopause = amenorrhea of more than 12 consecutive months)
* Uncontrolled psychotic state
* History of drug or alcohol intoxication requiring hospitalization within 12 months prior to randomization
* Recent or scheduled surgery within 6 months of randomization
* History of organ or hematopoietic marrow transplantation (except corneal transplantation performed at least 12 weeks prior to randomization)
* Primary or secondary immune deficiency
* Concomitant treatment with any of the following:

  * Methotrexate, leflunomide, cyclosporin A, azathioprine, mycophenolate mofetil, Janus kinase inhibitors, abatacept, secukinumab, anti-TNF-α, anakinra, ustekinumab, or any other immunosuppressive drug within 12 weeks prior to randomization
  * Rituximab or other anti-CD20 agent within 1 year prior to randomization
  * Cyclophosphamide in the year prior to randomization
* History of long-term corticosteroid therapy for conditions other than GCA or PPR. (NB: dermocorticoids, inhaled corticosteroids, and corticosteroid joint infiltrations are allowed during the study)
* Patient who has previously received ≥3 courses of oral corticosteroids for a disease other than GCA or RRP within 6 months prior to randomization
* Ongoing anti-tuberculosis treatment at the time of randomization
* Infections:

  * Current viral hepatitis B or C
  * Ongoing HIV infection
  * Severe infection requiring hospitalization within 30 days prior to randomization
* Any unstable or poorly controlled condition or disease, acute or chronic, not related to GCA, and considered a contraindication to tocilizumab therapy in the opinion of the investigator
* Neoplasia < 5 years, (except cervical cancer in situ and skin carcinoma, except melanoma, with R0 resection)

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
The relapse-free survival in both groups (immediate vs. gradual discontinuation) | at 26 weeks of follow-up
  The relapse-free survival in both groups (immediate vs. gradual discontinuation) defined as the time from S0 (start of immediate/progressive discontinuation strategy) to relapse or death (any cause), whichever occurs first.

SECONDARY OUTCOMES:
Relapse-free survival in both groups (immediate vs. gradual discontinuation) | at 26, 52 and 78 weeks of follow-up
Cumulative prednisone dose | at 26, 52 and 78 weeks of follow-up
Quality of life scores (HAQ) | at 0, 12, 26, 52 and 78 weeks of follow-up
FACIT-Fatigue score | at 0, 12, 26, 52 and 78 weeks of follow-up
Percentage of patients in remission without prednisone | at 26, 52 and 78 weeks of follow-up
Percentage of patients in remission with prednisone dose ≤5 mg/day | at 26, 52 and 78 weeks of follow-up
Frequency and type of adverse events in both groups | during the first 78 weeks after inclusion
Frequency of corticosteroid-related side effects (GTI score) in both groups | at baseline and at 52 weeks of follow-up
Quality of life scores (SF-36) | at 0, 12, 26, 52 and 78 weeks of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Derived] Samson M, Fournel I, Bourredjem A, Cortier M, Galizzi E, Cransac A, Cladiere C, Fleck C, Brayer M, Carpentier M, Alberini JL, Devilliers H, Bonnotte B. Immediate versus gradual TocilizuMab discontinuAtion in GIant Cell Arteritis: protocol of the multicentre randomised open-label MAGICA trial. BMJ Open. 2025 Oct 9;15(10):e108115. doi: 10.1136/bmjopen-2025-108115. PMID 41067765